CLINICAL TRIAL: NCT03183869
Title: Fecal Microbial Transplantation in Relapsing Multiple Sclerosis Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Primary Investigator passed away.
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MS-FMT-001
Record Dates: First submitted 2017-05-09; First posted 2017-06-12 (Actual); Results first posted 2019-12-02 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Autoimmune Diseases; Relapsing Multiple Sclerosis
Keywords: microbiome; multiple sclerosis; microbiota; gut
MeSH Terms: conditions — Autoimmune Diseases; Multiple Sclerosis | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: This is a prospective, cross-over, open label, randomized 1:1 early versus delayed groups, interventional [FMT] versus no interventional [no FMT] controlled trial to explore the effects of FMT from a healthy donor to RMS patients and investigate whether this can influence disease activity based on a panel of biological markers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Intervention (Active Comparator): Fecal microbiota via enema at Month 1, 2, 3. 4, 5 and month 6 along with stool, urine and blood collection. At months 7, 8, 9, 10, 11 and 12 only stool, urine and blood collection.
  Interventions: Drug: Fecal microbiota
- Late Intervention (Active Comparator): At months 1, 2, 3, 4, 5 and 6, stool, urine and blood collection. Fecal microbiota via enema at month 6, 7, 8, 9, 10, 11and 12 months along with stool, urine and blood collection.
  Interventions: Drug: Fecal microbiota

INTERVENTIONS:
Drug: Fecal microbiota — fecal microbial transplantation
  Other Names: fecal microbial transplantation

SUMMARY:
The proposed randomized, open label, with treat as usual control group (standard treatment or any disease modifying drugs), crossover phase II study will be conducted in 40 patients (n=20 per group) with the relapsing forms of multiple sclerosis according to the McDonald 2010 Criteria.

Patients will be randomized into 2 intervention groups. One will receive the FMT from month 1 and for the first 6 months (early intervention group). On the other hand, the other group will be a control group during the first 6 months and will receive the FMT for the last 6 months of the study. Patients will be screened for eligibility based on MS diagnosis and EDSS and if eligible then consented. All qualified patients will not be currently or recently treated with high dose steroids.

DETAILED DESCRIPTION:
At Visit 1, before FMT(fecal microbial transplantation), patients will be evaluated for their vital signs, medical history and concomitant medications. Also before transplantation, patient's stool will be collected to study their microbial profile, blood collected for analysis to evaluate cytokines levels as well as blood DNA bacteria and finally, urinalysis to assess gut permeability (baseline). Other assessments (prior to the first dose of therapy) include an Expanded Disability Status Scale (EDSS), pregnancy test (if applicable), physical exam and ECG. Blood samples are also taken at month 1 in order to establish a baseline for routine chemistry/hematology. After all these assessments FMT will be performed by a trained nurse via a rectal enema.

FMT for the early intervention group will be at V1, 2, 2.1, 2.2, V3 and V4. FMT randomized to late intervention group will be V4, 5, 6, 6.1.6.2, 6.3 and V7

Both groups, at Visit 1, Visit 4 and Visit 7, patients will be instructed to drink lactulose solution and collect the urine throughout the previous night and first thing in the morning. A proper collecting bottle will be provided and will also undergo a contrast-enhanced brain MRI scan at Robarts Institute London Ontario.

Those randomized to the Early Intervention group, will return to the clinic for visit 2, 1 month after the first FMT(fecal microbial transplantation). Another stool sample to evaluate the microbial before the second FMT will be collected and peripheral blood samples for cytokines and blood bacterial DNA analysis. Both groups this same routine procedure repeated at visits 2.1, 2.2, 3, 4, 5, 6, 6.1.6.2, 6.3 and visit 7. Another safety assessment 2 weeks after FMT is to review any adverse events that may have occurred.

Both groups will have an MRI at M1, M6 and M12.

ELIGIBILITY:
Inclusion Criteria:

* Have a confirmed diagnosis of relapsing MS defined by the 2010 Revised McDonald Criteria for the Diagnosis of Multiple Sclerosis
* Any disease duration will be accepted.
* Have a baseline EDSS of = or <7.0
* Older than 18 years of age.
* Be able to attend all clinic appointments without interruption
* Patients must be able to understand English sufficiently well to understand and comply with the clinic and medication schedules and procedures.
* Be willing and able to give written informed consent
* Negative blood pregnancy test at screening

Exclusion Criteria:

* Not meeting all of the above inclusion criteria
* Pregnancy or breastfeeding
* Current or recent [in the last 90 days] exposure to high dose corticosteroids
* Ongoing use of antibiotics
* Standard of care exclusions for MRI scans
* Presence of a chronic intestinal disease e.g. Celiac, malabsorption, colonic tumor
* Inability to provide informed written consent.
* Immunosuppression from transplantation, HIV, cancer chemotherapy or ongoing use of any immunosuppressive agents.
* Concomitant inflammatory diseases
* Pregnant women
* Any contra-indications for MRI. Participants are to be screened by a CMRTO (The College of Medical Radiation Technologists of Ontario) certified MRI Technologist in order to determine the MRI compatibility or exclusion of implantable/external devices according to the manufacturer's safety guidelines. The devises include cerebral aneurysm clips, neuro-stimulator, mechanical heart valves, cardiac stents, IUDs(intrauterine device), vena cava filters, shunts, embolization coils, cochlear implants, non-removable prosthesis/artificial limbs. Contraindications are pacemaker of defibrillator, shrapnel/metallic fragments, previous brain surgery, seizure, severe claustrophobia, weight or body index that will prevent a successful MRI study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-08-24 (Actual); Primary Completion 2018-11-19 (Actual); Study Completion 2019-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Kremenchutzky, MD, FRCP, Principal Investigator — London Health Science Centre
Locations (1):
- London Health Sciences Centre, University Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cantarel BL, Waubant E, Chehoud C, Kuczynski J, DeSantis TZ, Warrington J, Venkatesan A, Fraser CM, Mowry EM. Gut microbiota in multiple sclerosis: possible influence of immunomodulators. J Investig Med. 2015 Jun;63(5):729-34. doi: 10.1097/JIM.0000000000000192. PMID 25775034
- [Background] Miyake S, Kim S, Suda W, Oshima K, Nakamura M, Matsuoka T, Chihara N, Tomita A, Sato W, Kim SW, Morita H, Hattori M, Yamamura T. Dysbiosis in the Gut Microbiota of Patients with Multiple Sclerosis, with a Striking Depletion of Species Belonging to Clostridia XIVa and IV Clusters. PLoS One. 2015 Sep 14;10(9):e0137429. doi: 10.1371/journal.pone.0137429. eCollection 2015. PMID 26367776
- [Background] Tremlett H, Fadrosh DW, Faruqi AA, Hart J, Roalstad S, Graves J, Lynch S, Waubant E; US Network of Pediatric MS Centers. Gut microbiota composition and relapse risk in pediatric MS: A pilot study. J Neurol Sci. 2016 Apr 15;363:153-7. doi: 10.1016/j.jns.2016.02.042. Epub 2016 Feb 20. PMID 27000242
- [Background] Lavasani S, Dzhambazov B, Nouri M, Fak F, Buske S, Molin G, Thorlacius H, Alenfall J, Jeppsson B, Westrom B. A novel probiotic mixture exerts a therapeutic effect on experimental autoimmune encephalomyelitis mediated by IL-10 producing regulatory T cells. PLoS One. 2010 Feb 2;5(2):e9009. doi: 10.1371/journal.pone.0009009. PMID 20126401
- [Background] Kelly CR, de Leon L, Jasutkar N. Fecal microbiota transplantation for relapsing Clostridium difficile infection in 26 patients: methodology and results. J Clin Gastroenterol. 2012 Feb;46(2):145-9. doi: 10.1097/MCG.0b013e318234570b. PMID 22157239
- [Background] Kwon HK, Kim GC, Kim Y, Hwang W, Jash A, Sahoo A, Kim JE, Nam JH, Im SH. Amelioration of experimental autoimmune encephalomyelitis by probiotic mixture is mediated by a shift in T helper cell immune response. Clin Immunol. 2013 Mar;146(3):217-27. doi: 10.1016/j.clim.2013.01.001. Epub 2013 Jan 16. PMID 23416238
- [Background] Mielcarz DW, Kasper LH. The gut microbiome in multiple sclerosis. Curr Treat Options Neurol. 2015 Apr;17(4):344. doi: 10.1007/s11940-015-0344-7. PMID 25843302
- [Background] Hooper LV, Littman DR, Macpherson AJ. Interactions between the microbiota and the immune system. Science. 2012 Jun 8;336(6086):1268-73. doi: 10.1126/science.1223490. Epub 2012 Jun 6. PMID 22674334
- [Background] Wang S, Xu M, Wang W, Cao X, Piao M, Khan S, Yan F, Cao H, Wang B. Systematic Review: Adverse Events of Fecal Microbiota Transplantation. PLoS One. 2016 Aug 16;11(8):e0161174. doi: 10.1371/journal.pone.0161174. eCollection 2016. PMID 27529553

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Early Intervention | Late Intervention
Started | 4 | 7
Completed | 0 | 2
Not Completed | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Intervention | Late Intervention | Total
Number analyzed (Participants) | 4 | 7 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 6 | 10
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 1 | 2 | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Effect of Fecal Microbial Transplantation in Peripheral Blood Cytokines Within Relapsing Multiple Sclerosis Patients
Description: Luminex test to evaluate the levels of 25 cytokines in peripheral blood pre-fecal transplant and post fecal transplant. Due to early termination of the trial, we didn't meet the number of participants required for statistical analysis; therefore, we analyzed the data pre and post FMT, rather than early and late intervention groups as originally planned. Due to the small sample size there was a large variation between cytokine levels of each participant for pre and post FMT, resulting in large standard deviations.
Time Frame: Within 6 months
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Pre-FMT: Cytokine values before fecal microbial transplants.
  Fecal microbiota: fecal microbial transplantation
- Post-FMT: Cytokine values after fecal microbial transplants.
  Fecal microbiota: fecal microbial transplantation
Arm/Group | Pre-FMT | Post-FMT
Number analyzed (Participants) | 10 | 10
ng/mL
  IL17F | 0.082 (0.076) | 0.093 (0.148)
  GM-CSF | 0.171 (0.186) | 0.261 (0.524)
  IFN Gamma | 0.064 (0.046) | 0.078 (0.070)
  IL-10 | 0.026 (0.024) | 0.024 (0.026)
  MIP3 Alpha | 0.049 (0.035) | 0.036 (0.023)
  IL-12p70 | 0.026 (0.019) | 0.033 (0.043)
  IL-13 | 0.091 (0.186) | 0.084 (0.181)
  IL-15 | 0.030 (0.038) | 0.036 (0.054)
  IL-17a | 0.018 (0.018) | 0.023 (0.039)
  IL-22 | 0.414 (0.443) | 0.559 (0.811)
  IL-9 | 0.036 (0.039) | 0.031 (0.042)
  IL-1 Beta | 0.013 (0.011) | 0.013 (0.013)
  IL-33 | 0.123 (0.097) | 0.086 (0.114)
  IL-2 | 0.016 (0.017) | 0.016 (0.024)
  IL-21 | 0.042 (0.031) | 0.040 (0.043)
  IL-4 | 0.428 (0.426) | 0.425 (0.380)
  IL-23 | 8.778 (8.549) | 10.906 (16.971)
  IL-5 | 0.023 (0.021) | 0.028 (0.026)
  IL-6 | 0.055 (0.117) | 0.056 (0.129)
  IL-17E | 0.149 (0.153) | 0.203 (0.342)
  IL-27 | 1.534 (0.795) | 1.792 (1.322)
  IL-31 | 0.156 (0.220) | 0.198 (0.280)
  TNF alpha | 0.042 (0.033) | 0.053 (0.036)
  TNF beta | 0.313 (0.585) | 0.306 (0.627)
  IL-28a | 1.190 (2.512) | 1.704 (2.499)

2. Secondary Outcome: Evaluate Effect of Fecal Microbial Transplantation in Gut Microbiome
Description: PCR (polymerase chain reaction) to assess blood DNA bacteria
Time Frame: Monthly for 6 months
Reporting Status: Not Posted

3. Secondary Outcome: Evaluate Effect of Fecal Microbial Transplantation in Gut Permeability
Description: Urinalysis to evaluate lactulose and mannitol levels
Time Frame: Baseline, 6 months, 12 months
Reporting Status: Not Posted

4. Secondary Outcome: Evaluate Treatment Clinical Safety: Neurological Exam Using the Expanded Disability Status Scale
Description: Neurological exam using the Expanded Disability Status Scale
Time Frame: Monthly for 6 months
Reporting Status: Not Posted

5. Secondary Outcome: Evaluate Treatment Safety: MRI to Access Subclinical Disease Activity
Description: MRI to access subclinical disease activity
Time Frame: Baseline, 6 months and 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year - Nov2017 - Nov2018
Arm/Group | Early Intervention | Late Intervention
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/7
Other Adverse Events (participants affected / at risk) | 3/4 | 5/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Early Intervention (N=4) | Late Intervention (N=7)
Nausea (Gastrointestinal disorders) | 3 | 0
Hives (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Cardiac disorders) | 0 | 1
Difficulty Swallowing (Gastrointestinal disorders) | 0 | 1
Vaginal Yeast Infection (Reproductive system and breast disorders) | 0 | 1
Ear Infection (Ear and labyrinth disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-09): https://cdn.clinicaltrials.gov/large-docs/69/NCT03183869/Prot_SAP_000.pdf